CLINICAL TRIAL: NCT02027883
Title: Comparison of Ventricular Fibrillation Induction Techniques During Medtronic Implantable Cardioverter Defibrillator Implant
Brief Title: Comparison of VF Induction Techniques During Medtronic ICD Implant (VF) (ICD)
Acronym: VF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James Merrill (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, James Merrill, James Merrill, MD, FACC, Wellmont CVA Heart Institute
Organization: Wellmont CVA Heart Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VF Induction
Record Dates: First submitted 2013-12-31; First posted 2014-01-06 (Estimated); Results first posted 2014-12-30 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-04

CONDITIONS: Cardiomyopathy
Keywords: Defibrillators; Ventricular Fibrillation Induction Testing
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nominal Parameter (Active Comparator): Nominal T shock setting
  Interventions: Device: Nominal T shock setting
- Experimental Parameter (Experimental): Educated T shock setting
  Interventions: Device: Educated T shock setting

INTERVENTIONS:
Device: Nominal T shock setting — Nominal Parameter Set 1 Programming Values for EnTrust
  Other Names: Medtronic ICDs
  Arms: Nominal Parameter
Device: Educated T shock setting — Experimental Parameter Set 2 Programming Values
  Other Names: Medtronic ICDs
  Arms: Experimental Parameter

SUMMARY:
As the indications for Implantable Cardioverter Defibrillator implantation expand, minimizing implant time is critical. Also, patients receiving biventricular ICDs are sometimes more unstable and minimization of sedation time is crucial. Multiple induction attempts, with a 1-Joule shock, can cause disruption in lead position. Therefore limiting the number of attempts will allow for better lead stability throughout the procedure and a more straightforward implant process.

Investigator proposes a detailed documentation of success rates from various Ventriculart Fibrillation induction methods during implant of Medtronic defibrillation capable devices.

DETAILED DESCRIPTION:
Our clinical experience has found that attempts to induce patients receiving ICDs at implant using the nominal Medtronic T-shock settings are not always effective at inducing ventricular fibrillation. When this results, a change to the parameters for T-shock is made before reattempting to induce ventricular fibrillation in patients undergoing ICD implantation.

Another available induction method is 50 Hz Burst. "The 50 Hz Burst induction is designed to induce VF by delivering a rapid burst of pacing pulses. The amplitude and pulse width of these pulses are selectable, but the pacing interval is fixed at 20 ms."2 If multiple attempts using the T-shock method are unsuccessful, 50 Hz Burst provides an additional method for inducing ventricular fibrillation. It is a less desirable method since it can result in very fine VF that is difficult to identify the initiation of possibly resulting in longer times in VF causing higher defibrillation threshold or in undersensing due to the fine nature of the rhythm.

T-shock has been found to be a fast and reliable method for inducing ventricular fibrillation in ICD implants. Greater success of inducing ventricular fibrillation using the T-shock method has been found when the energy of the T-shock was higher and the coupling interval was shorter. In addition, increasing the shock strength increases the window of vulnerability. For the T-shock method to be most efficient, initial success at inducing ventricular fibrillation, and therefore a reduced number of attempts, is important. This requires a better understanding of the optimal programmed settings for the initial T-shock induction attempt.

Moreover, in recent years, ICD indications have grown to include primary prevention patients. These patients may have different vulnerable periods than patients previously evaluated to develop Medtronic nominal settings.

Our clinical experience has found that the nominal T-shock settings are only effective at inducing ventricular fibrillation approximately seventy-five percent of the time. However, a detailed collection of success rates has not been performed.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing Medtronic ICD or Cardiac Resynchronization Therapy-Defibrillator implant (initial implant or generator replacement) will be included.

Exclusion Criteria:

* Any patient who is medically unstable and testing is deemed unsafe by physician will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wellmont CVA Heart Institute, Kingsport, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bardy G, Mehra R, Johnson G, Kudenchuk P, Dolack G, Poole J, Hofer B: Low energy pulsing on the T-wave: A new programming method for intentional, device mediated induction of ventricular fibrillation for defibrillation testing. PACE 15(4, Pt II): 562, 1992.
- [Background] Bhandari AK, Isber N, Estioko M, Ziccardi T, Cannom DS, Park Y, Lerman RD, Prejean C, Sun GW. Efficacy of low-energy T wave shocks for induction of ventricular fibrillation in patients with implantable cardioverter defibrillators. J Electrocardiol. 1998 Jan;31(1):31-7. doi: 10.1016/s0022-0736(98)90004-8. PMID 9533375
- [Background] Marquis DR Reference Manual, Medtronic, Inc.
- [Background] Mitchell L, Yee R, Talajic M, Newman D, Sheldon R, Kerr C, Kus T, Boyle A, Canadian Jewel PCD Investigators: Low-energy, T-wave synchronous, interval shock for rapid, reliable ventricular fibrillation induction by an implantable cardioverter defibrllattor. PACE, 17(4, Pt II): 851, 1994.
- [Background] Swartz J, Stanton M, DeGroot P, Mehra R: Influence of T-wave shock energy on ventricular fibrillation vulnerability in humans. JACC 1995 Conference Abstracts: 214A, 1995.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nominal Parameter | Experimental Parameter
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nominal Parameter | Experimental Parameter | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 18 | 45
  >=65 years | 23 | 32 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.82 (13.68403) | 66.68 (10.51809) | 64.25 (12.38554)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 38 | 40 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 50 | 50 | 100
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 50 | 50 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100
VF Induction amount of participants [Number; unit: participants] — Number of subjects that participated in the VF induction study protocol.
  participants | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Sustained Ventricular Fibrillation
Description: The primary endpoint is the successful induction of sustained ventricular fibrillation.
Time Frame: 2 hours
Measure: Number; unit: participants
Arm/Group | Nominal Parameter | Experimental Parameter
Number analyzed (Participants) | 50 | 50
participants | 38 | 35

2. Secondary Outcome: Factors
Description: Determine if any pre-implant patient demographics are factors impacting T-shock success according to parameter settings.
Time Frame: 2 hours
Measure: Number; unit: participants
Arm/Group | Nominal Parameter | Experimental Parameter
Number analyzed (Participants) | 50 | 50
participants
  Successful Male Participants | 30 | 28
  Successful Female participants | 8 | 7
  Unsuccessful Male Participants | 8 | 12
  Unsuccessful Female Participants | 4 | 3

3. Other Pre Specified Outcome: Safety Monitoring
Description: Number of participants that were monitored for safety issues, including increased heart rate, blood pressure, decreased oximetry levels, and stable rhythm during the entire procedure.
Time Frame: 2 hours
Measure: Number; unit: participants
Groups:
- Nominal Parameter: Nominal T shock setting
  Nominal T shock setting: Nominal Parameter Set 1 Programming Values for EnTrust
  The standard T-Shock method was successful in 76% of the patients. 38 out of 50 patients Ventricular Fibrillation was induced with the nominal T shock method. In contrast, 87 % or 13 out of 15 that failed to induce Ventricular Fibrillation using the educated T-Shock method was successfully induced when crossed to the nominal T-shock method.
- Experimental Parameter: Educated T shock setting
  Educated T shock setting: Experimental Parameter Set 2 Programming Values
  The educated T shock setting method was successful in 70% of the patients. 35 out of 50 patients Ventricular Fibrillation was induced with the educated T- shock method. Of the 12 patients that were did not have Ventricular fibrillation induced with the nominal T-shock method, they were all successfully induced with the educated T-Shock method.
Arm/Group | Nominal Parameter | Experimental Parameter
Number analyzed (Participants) | 50 | 50
participants | 50 | 50

ADVERSE EVENTS:
Time Frame: The patient's were observed for adverse events from the time of consent to the time they met the primary endpoint.
Arm/Group | Nominal Parameter | Experimental Parameter
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other